CLINICAL TRIAL: NCT05383209
Title: A Phase 2, Multicenter, Prospective, Double-masked, Parallel Study of EYP-1901, a Tyrosine Kinase Inhibitor (TKI), Compared to Sham for the Improvement of Moderately Severe to Severe Nonproliferative Diabetic Retinopathy (NPDR)
Brief Title: Study of EYP-1901 in Patients With Nonproliferative Diabetic Retinopathy (NPDR)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EyePoint Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EYP-1901-204
Record Dates: First submitted 2022-05-10; First posted 2022-05-20 (Actual); Results first posted 2025-07-28 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Nonproliferative Diabetic Retinopathy
Keywords: NPDR; EYP-1901; EyePoint
MeSH Terms: interventions — vorolanib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- EYP-1901 2060 ug (Experimental): EYP-1901 2060 ug; single injection
  Interventions: Drug: EYP-1901
- EYP-1901 3090 ug (Experimental): EYP-1901 3090 ug; single injection
  Interventions: Drug: EYP-1901
- Sham IVT (Sham Comparator): Sham IVT; single injection
  Interventions: Other: Sham IVT

INTERVENTIONS:
Drug: EYP-1901 — EYP-1901 will be administered to the study eye by a single injection through the pars plana using a pre-loaded applicator with a 22-gauge needle. Each EYP-1901 IVT insert has been designed to deliver vorolanib into the vitreous humor for approximately 6 to 9 months.
  Other Names: Vorolanib
  Arms: EYP-1901 2060 ug; EYP-1901 3090 ug
Other: Sham IVT — Sham injections will be used to maintain masking of investigational EYP-1901 therapy for study subjects.
  Arms: Sham IVT

SUMMARY:
A prospective, randomized, double-masked study that evaluated the ocular efficacy and safety of two doses of the EYP-1901 intravitreal (IVT) insert compared to sham.

DETAILED DESCRIPTION:
This study evaluated the ocular efficacy and safety of two doses of the EYP-1901 IVT insert compared to sham using a randomized double-masked trial design.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a hemoglobin A1c <=12%
* Study eye with moderately severe to severe Non proliferative Diabetic Retinopathy (NPDR) (based on the Diabetic Retinopathy Severity Scale (DRSS) levels 47 or 53)
* Best corrected visual acuity (BCVA) using Early Treatment Diabetic Retinopathy Study (ETDRS) letter score in the study eye of >=69 letters (approximate Snellen equivalent of 20/40 or better).

Exclusion Criteria:

* Presence of any active Center involved-diabetic macular edema in the study eye as determined by the Investigator on clinical examination, or within the central subfield thickness (CST) of the study eye, with a CST threshold greater than 320 microns.
* Any evidence or documented history of prior focal or grid laser photocoagulation or any pan-retinal photocoagulation (PRP) in the study eye in the last 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2022-09-28 (Actual); Primary Completion 2024-02-12 (Actual); Study Completion 2024-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramiro Ribeiro, MD, PhD, Study Director — EyePoint Pharmaceuticals
Locations (36):
- United States (36):
  - EyePoint Investigative Site, Phoenix, Arizona
  - EyePoint Investigative Site, Huntington Beach, California
  - EyePoint Investigative Site, Oxnard, California
  - EyePoint Investigative Site, Palm Desert, California
  - EyePoint Investigative Site, Pasadena, California
  - EyePoint Investigative Site, Poway, California
  - EyePoint Investigative Site, Sacramento, California
  - EyePoint Investigative Site, Danbury, Connecticut
  - EyePoint Investigative Site, Clearwater, Florida
  - EyePoint Investigative Site, Melbourne, Florida
  - EyePoint Investigative Site, Miami, Florida
  - EyePoint Investigative Site, Winter Haven, Florida
  - EyePoint Investigative Site, Lemont, Illinois
  - EyePoint Investigative Site, Indianapolis, Indiana
  - EyePoint Investigative Site, Lenexa, Kansas
  - EyePoint Investigative Site, Baltimore, Maryland
  - EyePoint Investigative Site, Hagerstown, Maryland
  - EyePoint Investigative Site, Springfield, Massachusetts
  - EyePoint Investigative Site, Reno, Nevada
  - EyePoint Investigative Site, Bloomfield, New Jersey
  - EyePoint Investigative Site, Toms River, New Jersey
  - EyePoint Investigative Site, Great Neck, New York
  - EyePoint Investigative Site, Erie, Pennsylvania
  - EyePoint Investigative Site, Florence, South Carolina
  - EyePoint Investigative Site, Ladson, South Carolina
  - EyePoint Investigative Site, Rapid City, South Dakota
  - EyePoint Investigative Site, Germantown, Tennessee
  - EyePoint Investigative Site, Abilene, Texas
  - EyePoint Investigative Site, Austin, Texas
  - EyePoint Investigative Site, Houston, Texas
  - EyePoint Investigative Site, McAllen, Texas
  - EyePoint Investigative Site, Plano, Texas
  - EyePoint Investigative Site, San Antonio, Texas
  - EyePoint Investigative Site, The Woodlands, Texas
  - EyePoint Investigative Site, Lynchburg, Virginia
  - EyePoint Investigative Site, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase 2 prospective, randomized, double-masked study was conducted in adult subjects with NPDR at 25 sites in the United States between 28 September 2022 and 06 May 2024.
Pre-assignment Details: This study consists of a screening period (up to 30 days) and treatment period (48 weeks). A total of 77 subjects were enrolled in the study.
Groups:
- Sham Injection: Subjects received a single dose of sham IVT injection on Day 1.
- EYP-1901 2060 mcg: Subjects received a single dose of EYP-1901 2060 microgram (mcg) IVT injection on Day 1.
- EYP-1901 3090 mcg: Subjects received a single dose of EYP-1901 3090 mcg IVT injection on Day 1.
Period: Overall Study
Arm/Group | Sham Injection | EYP-1901 2060 mcg | EYP-1901 3090 mcg
Started | 26 | 26 | 25
Completed | 21 | 23 | 20
Not Completed | 5 | 3 | 5
Not completed — Adverse Event: Non-ocular | 0 | 1 | 0
Not completed — Lost to Follow-up | 2 | 1 | 4
Not completed — Withdrawal by Subject | 2 | 0 | 1
Not completed — Death | 1 | 0 | 0
Not completed — Other | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all subjects who received at least 1 dose of study treatment (EYP-1901 or sham).
Groups:
- EYP-1901 2060 mcg: Subjects received a single dose of EYP-1901 2060 mcg IVT injection on Day 1.
- Total: Total of all reporting groups
Arm/Group | Sham Injection | EYP-1901 2060 mcg | EYP-1901 3090 mcg | Total
Number analyzed (Participants) | 26 | 26 | 25 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (11.95) | 56.8 (11.79) | 60.2 (9.98) | 57.9 (11.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 9 | 34
  Male | 13 | 14 | 16 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 8 | 8 | 25
  Not Hispanic or Latino | 17 | 16 | 17 | 50
  Unknown or Not Reported | 0 | 2 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 1 | 1 | 4
  Black | 1 | 3 | 5 | 9
  White | 21 | 19 | 18 | 58
  American Indian or Alaskan Native | 0 | 2 | 0 | 2
  Other | 2 | 1 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Improved >=2 Steps From Baseline in the DRSS Score at Week 36
Description: The DRSS used to describe overall retinopathy severity as well as the change in severity over time in the study eye. Severity ranges from level 10 (diabetic retinopathy absent) to level 85 (advanced proliferative diabetic retinopathy (PDR): posterior fundus obscured, or center of macula detached). Here, DRSS describes severity level 47 (moderately severe NPDR) and level 53 (severe NPDR) at Week 36 from baseline.
Time Frame: Baseline (Day 1) and Week 36
Population: The FAS included all subjects who received at least 1 dose of study treatment (EYP-1901 or sham).
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Sham Injection | EYP-1901 2060 mcg | EYP-1901 3090 mcg
Number analyzed (Participants) | 20 | 20 | 21
percentage of subjects | 5.0 [0.1 to 24.9] | 0 [0.0 to 16.8] | 4.8 [0.1 to 23.8]
Statistical Analysis 1: Comparison: Sham Injection vs EYP-1901 2060 mcg; Test type: Other; Difference in response percentage = -5.0, 95% CI 2-sided [-24.9 to 13.4]
Statistical Analysis 2: Comparison: Sham Injection vs EYP-1901 3090 mcg; Test type: Other; Slope = -0.2, 95% CI 2-sided [-20.6 to 20.6]

2. Secondary Outcome: Percentage of Subjects Improved >=2 Steps From Baseline in the DRSS Score at Week 24 and Week 48
Description: The DRSS used to describe overall retinopathy severity as well as the change in severity over time in the study eye. Severity ranges from level 10 (diabetic retinopathy absent) to level 85 (advanced proliferative diabetic retinopathy (PDR): posterior fundus obscured, or center of macula detached). Here, DRSS describes severity levels 47 (moderately severe NPDR) and 53 (severe NPDR) at Weeks 24 and 48 from baseline.
Time Frame: Baseline (Day 1), Week 24, and Week 48
Population: The FAS included all subjects who received at least 1 dose of study treatment (EYP-1901 or sham).
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Groups:
- Sham Injection (Week 24); Sham Injection (Week 48): Subjects received a single dose of sham IVT injection on Day 1.
- EYP-1901 2060 mcg (Week 24); EYP-1901 2060 mcg (Week 48): Subjects received a single dose of EYP-1901 2060 mcg IVT injection on Day 1.
- EYP-1901 3090 mcg (Week 24); EYP-1901 3090 mcg (Week 48): Subjects received a single dose of EYP-1901 3090 mcg IVT injection on Day 1.
Arm/Group | Sham Injection (Week 24) | Sham Injection (Week 48) | EYP-1901 2060 mcg (Week 24) | EYP-1901 2060 mcg (Week 48) | EYP-1901 3090 mcg (Week 24) | EYP-1901 3090 mcg (Week 48)
Number analyzed (Participants) | 18 | 19 | 16 | 20 | 19 | 19
percentage of subjects | 0 [0.0 to 18.5] | 0 [0.0 to 17.6] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 17.6] | 5.3 [0.1 to 26.0]
Statistical Analysis 1: Comparison: EYP-1901 3090 mcg (Week 48); Test type: Other; Difference in response percentage = 5.3, 95% CI 2-sided [-13.2 to 26.0]

3. Secondary Outcome: Percentage of Subjects Improved >=2 Steps and >=3 Steps From Baseline in DRSS Score at Weeks 24, 36 and 48
Description: The DRSS used to describe overall retinopathy severity as well as the change in severity over time in the study eye. Severity ranges from level 10 (diabetic retinopathy absent) to level 85 (advanced PDR: posterior fundus obscured, or center of macula detached). Here, DRSS describes severity level 47 (moderately severe NPDR) and level 53 (severe NPDR) at Weeks 24, 36 and 48 from baseline.
Time Frame: Baseline (Day 1) and Weeks 24, 36 and 48
Population: The FAS included all subjects who received at least 1 dose of study treatment (EYP-1901 or sham). Only subjects analyzed at specific timepoints are reported.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Sham Injection | EYP-1901 2060 mcg | EYP-1901 3090 mcg
Number analyzed (Participants) | 26 | 26 | 25
percentage of subjects
  >=2-step improvement in DRSS: Week 24: number analyzed (Participants) | 18 | 16 | 19
  >=2-step improvement in DRSS: Week 24 | 0 [0.0 to 18.5] | 0 [0.0 to 20.6] | 0 [0.0 to 17.6]
  >=2-step improvement in DRSS: Week 36: number analyzed (Participants) | 20 | 20 | 21
  >=2-step improvement in DRSS: Week 36 | 5.0 [0.1 to 24.9] | 0 [0.0 to 16.8] | 4.8 [0.1 to 23.8]
  >=2-step improvement in DRSS: Week 48: number analyzed (Participants) | 19 | 20 | 19
  >=2-step improvement in DRSS: Week 48 | 0 [0.0 to 17.6] | 0 [0.0 to 16.8] | 5.3 [0.1 to 26.0]
  >=3-step improvement in DRSS: Week 24: number analyzed (Participants) | 18 | 16 | 19
  >=3-step improvement in DRSS: Week 24 | 0 [0.0 to 18.5] | 0 [0.0 to 20.6] | 0 [0.0 to 17.6]
  >=3-step improvement in DRSS: Week 36: number analyzed (Participants) | 20 | 20 | 21
  >=3-step improvement in DRSS: Week 36 | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.1]
  >=3-step improvement in DRSS: Week 48: number analyzed (Participants) | 19 | 20 | 19
  >=3-step improvement in DRSS: Week 48 | 0 [0.0 to 17.6] | 0 [0.0 to 16.8] | 0 [0.0 to 17.6]

4. Secondary Outcome: Percentage of Subjects Worsened >=2 Steps and >=3 Steps From Baseline in DRSS Score at Weeks 24, 36 and 48
Description: as for outcome 3
Time Frame: Baseline (Day 1) and Weeks 24, 36 and 48
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Sham Injection | EYP-1901 2060 mcg | EYP-1901 3090 mcg
Number analyzed (Participants) | 26 | 26 | 25
percentage of subjects
  >=2-step worsening in DRSS: Week 24: number analyzed (Participants) | 18 | 16 | 19
  >=2-step worsening in DRSS: Week 24 | 0 [0.0 to 18.5] | 6.3 [0.2 to 30.2] | 0 [0.0 to 17.6]
  >=2-step worsening in DRSS: Week 36: number analyzed (Participants) | 20 | 20 | 21
  >=2-step worsening in DRSS: Week 36 | 10.0 [1.2 to 31.7] | 5.0 [0.1 to 24.9] | 0 [0.0 to 16.1]
  >=2-step worsening in DRSS: Week 48: number analyzed (Participants) | 19 | 20 | 19
  >=2-step worsening in DRSS: Week 48 | 0 [0.0 to 17.6] | 5.0 [0.1 to 24.9] | 0 [0.0 to 17.6]
  >=3-step worsening in DRSS: Week 24: number analyzed (Participants) | 18 | 16 | 19
  >=3-step worsening in DRSS: Week 24 | 0 [0.0 to 18.5] | 0 [0.0 to 20.6] | 0 [0.0 to 17.6]
  >=3-step worsening in DRSS: Week 36: number analyzed (Participants) | 20 | 20 | 21
  >=3-step worsening in DRSS: Week 36 | 5.0 [0.1 to 24.9] | 0 [0.0 to 16.8] | 0 [0.0 to 16.1]
  >=3-step worsening in DRSS: Week 48: number analyzed (Participants) | 19 | 20 | 19
  >=3-step worsening in DRSS: Week 48 | 0 [0.0 to 17.6] | 0 [0.0 to 16.8] | 0 [0.0 to 17.6]

5. Secondary Outcome: Percentage of Subjects Who Developed a Vision-Threatening Complication Due to Diabetic Retinopathy at Weeks 24, 36 and 48
Description: The vision threatening complications in the study eye due to diabetic retinopathy were indicated by the presence of "Vitreous hemorrhage" or the presence of "Tractional retinal detachment" reported on the Ocular Examination - Dilated Ophthalmoscopy CRF (PDR events), and "Neovascularization for the Iris" answered as "Yes" or "Neovascularization for the Angle" answered as "Yes" per the Ocular Examination - Slit Lamp Biomicroscopy CRF (anterior segment neovascularization (ASNV) events).
Time Frame: Weeks 24, 36 and 48
Population: The FAS included all subjects who received at least 1 dose of study treatment (EYP-1901 or sham).
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Sham Injection | EYP-1901 2060 mcg | EYP-1901 3090 mcg
Number analyzed (Participants) | 26 | 26 | 25
percentage of subjects
  Week 24 | 0 [0.0 to 13.2] | 3.8 [0.1 to 19.6] | 0 [0.0 to 13.7]
  Week 36 | 3.8 [0.1 to 19.6] | 3.8 [0.1 to 19.6] | 0 [0.0 to 13.7]
  Week 48 | 3.8 [0.1 to 19.6] | 3.8 [0.1 to 19.6] | 0 [0.0 to 13.7]

6. Secondary Outcome: Percentage of Subjects Who Developed Center Involved-Diabetic Macular Edema (CI-DME) at Weeks 24, 36 and 48
Description: The CI-DME in the study eye occurred when a treatment emergent adverse event (TEAE) with a mapped preferred term of 'Cystoid macular oedema', 'Diabetic retinal oedema', or 'Macular oedema' occurred in the study eye, in combination with the temporally closest centrally read custom algorithm CST measurement being greater than or equal to 320 microns.
Time Frame: Weeks 24, 36 and 48
Population: The FAS included all subjects who received at least 1 dose of study treatment (EYP-1901 or sham).
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Sham Injection | EYP-1901 2060 mcg | EYP-1901 3090 mcg
Number analyzed (Participants) | 26 | 26 | 25
percentage of subjects
  Week 24 | 0 [0.0 to 13.2] | 0 [0.0 to 13.2] | 0 [0.0 to 13.7]
  Week 36 | 0 [0.0 to 13.2] | 0 [0.0 to 13.2] | 4.0 [0.1 to 20.4]
  Week 48 | 3.8 [0.1 to 19.6] | 0 [0.0 to 13.2] | 8.0 [1.0 to 26.0]

7. Secondary Outcome: Time to Develop Any Neovascular Vision Threatening Complication (PDR/ASNV) at Weeks 24, 36 and 48
Description: Time to develop any PDR/ASNV was computed as the date of the first development of PDR/ASNV in the study eye minus the date of study treatment administration plus 1 day, divided by 7 days per week.
Time Frame: Weeks 24, 36 and 48
Population: The FAS included all subjects who received at least 1 dose of study treatment (EYP-1901 or sham). Only subjects developed any PDR/ASNV at specific timepoint are analyzed.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Sham Injection | EYP-1901 2060 mcg | EYP-1901 3090 mcg
Number analyzed (Participants) | 26 | 26 | 25
weeks
  Week 24: number analyzed (Participants) | 0 | 1 | 0
  Week 24 |  | NA [NA to NA] — Median and 95% confidence interval data were not calculable due to no/low occurrence of PDR/ASNV events. |
  Week 36: number analyzed (Participants) | 1 | 1 | 0
  Week 36 | NA [NA to NA] — Median and 95% confidence interval data were not calculable due to no/low occurrence of PDR/ASNV events. | NA [NA to NA] — Median and 95% confidence interval data were not calculable due to no/low occurrence of PDR/ASNV events. |
  Week 48: number analyzed (Participants) | 1 | 1 | 0
  Week 48 | NA [NA to NA] — Median and 95% confidence interval data were not calculable due to no/low occurrence of PDR/ASNV events. | NA [NA to NA] — Median and 95% confidence interval data were not calculable due to no/low occurrence of PDR/ASNV events. |

8. Secondary Outcome: Time to Develop CI-DME Through Weeks 24, 36 and 48
Description: The occurrence of a CI-DME event in the study eye was identified via examination of centrally read custom algorithm CST data and adverse events.
Time Frame: Weeks 24, 36 and 48
Population: The FAS included all subjects who received at least 1 dose of study treatment (EYP-1901 or sham). Only subjects developed CI-DME event at specific timepoint are analyzed.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Sham Injection | EYP-1901 2060 mcg | EYP-1901 3090 mcg
Number analyzed (Participants) | 26 | 26 | 25
weeks
  Week 24: number analyzed (Participants) | 0 | 0 | 0
  Week 36: number analyzed (Participants) | 0 | 0 | 1
  Week 36 |  |  | NA [NA to NA] — Median and 95% confidence interval data were not calculable due to no/low occurrence of CI-DME events.
  Week 48: number analyzed (Participants) | 1 | 0 | 2
  Week 48 | NA [NA to NA] — Median and 95% confidence interval data were not calculable due to no/low occurrence of CI-DME events. |  | NA [NA to NA] — Median and 95% confidence interval data were not calculable due to no/low occurrence of CI-DME events.

9. Secondary Outcome: Percentage of Subjects Who Received Anti-Vascular Endothelial Growth Factor (VEGF) or Additional Standard of Care Intervention Due to Ocular Diabetic Complications at Weeks 24, 36 and 48
Description: Percentage of subjects who received anti-VEGF or additional standard of care intervention due to ocular diabetic complications in the study eye are reported. Anti-VEGF use was identified in reported concomitant medication data.
Time Frame: Weeks 24, 36 and 48
Population: The FAS included all subjects who received at least 1 dose of study treatment (EYP-1901 or sham).
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Sham Injection | EYP-1901 2060 mcg | EYP-1901 3090 mcg
Number analyzed (Participants) | 26 | 26 | 25
percentage of subjects
  Week 24 | 7.7 [0.9 to 25.1] | 7.7 [0.9 to 25.1] | 4.0 [0.1 to 20.4]
  Week 36 | 7.7 [0.9 to 25.1] | 7.7 [0.9 to 25.1] | 8.0 [1.0 to 26.0]
  Week 48 | 7.7 [0.9 to 25.1] | 7.7 [0.9 to 25.1] | 12.0 [2.5 to 31.2]

10. Secondary Outcome: Percentage of Subjects Who Received PRP at Weeks 24, 36 and 48
Description: Percentage of subjects who received PRP in the study eye, inclusive of subjects undergoing vitrectomy with endo-laser are reported.
Time Frame: Weeks 24, 36 and 48
Population: The FAS included all subjects who received at least 1 dose of study treatment (EYP-1901 or sham).
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Sham Injection | EYP-1901 2060 mcg | EYP-1901 3090 mcg
Number analyzed (Participants) | 26 | 26 | 25
percentage of subjects
  Week 24 | 0 [0.0 to 13.2] | 3.8 [0.1 to 19.6] | 0 [0.0 to 13.7]
  Week 36 | 0 [0.0 to 13.2] | 3.8 [0.1 to 19.6] | 0 [0.0 to 13.7]
  Week 48 | 0 [0.0 to 13.2] | 3.8 [0.1 to 19.6] | 0 [0.0 to 13.7]

11. Secondary Outcome: Area Under the Curve (AUC) for Change From Baseline in BCVA at Weeks 24, 36 and 48
Description: The AUC for change from baseline in BCVA in the study eye were summarized. The AUC through each time point of interest was computed using the trapezoidal rule normalized to months, with a final unit of letters.
Time Frame: Weeks 24, 36 and 48
Population: The FAS included all subjects who received at least 1 dose of study treatment (EYP-1901 or sham).
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Sham Injection | EYP-1901 2060 mcg | EYP-1901 3090 mcg
Number analyzed (Participants) | 26 | 26 | 25
letters
  Week 24: number analyzed (Participants) | 22 | 22 | 23
  Week 24 | -0.32 (2.969) | -1.58 (8.411) | 0.46 (4.070)
  Week 36: number analyzed (Participants) | 23 | 23 | 23
  Week 36 | -0.23 (3.234) | -1.52 (6.819) | 0.03 (4.562)
  Week 48: number analyzed (Participants) | 21 | 23 | 20
  Week 48 | -0.38 (3.127) | -1.44 (6.369) | -0.02 (5.311)

12. Secondary Outcome: Plasma Concentration of EYP-1901 and X-297 at Weeks 24, 36 and 48
Description: Blood samples were collected at the specific visits for the Pharmacokinetic (PK) analysis of EYP-1901 and its main metabolite concentrations.
Time Frame: Weeks 24, 36 and 48
Population: The PK analysis set included all subjects in the Safety set for whom at least 1 evaluable PK sample was available. Only subjects analysis at specific timepoints are reported.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | EYP-1901 2060 mcg | EYP-1901 3090 mcg
Number analyzed (Participants) | 26 | 25
mcg/mL
  EYP-1901: Week 24: number analyzed (Participants) | 22 | 21
  EYP-1901: Week 24 | 11.852 (5.6180) | 14.064 (5.0654)
  EYP-1901: Week 36: number analyzed (Participants) | 22 | 22
  EYP-1901: Week 36 | 7.660 (4.8187) | 9.708 (5.5782)
  EYP-1901: Week 48: number analyzed (Participants) | 23 | 19
  EYP-1901: Week 48 | 6.698 (3.7642) | 8.194 (3.5894)
  X-297: Week 24: number analyzed (Participants) | 22 | 21
  X-297: Week 24 | 0.000 (0.0000) | 0.000 (0.0000)
  X-297: Week 36: number analyzed (Participants) | 23 | 22
  X-297: Week 36 | 0.999 (4.7917) | 0.275 (1.2877)
  X-297: Week 48: number analyzed (Participants) | 23 | 19
  X-297: Week 48 | 0.000 (0.0000) | 0.657 (2.8631)

13. Secondary Outcome: Number of Subjects With Ocular and Non-Ocular TEAEs and Serious TEAEs up to Week 48
Description: An adverse event (AE) is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a patient or clinical investigation subject administered an investigational or marketed (medicinal) product and that does not necessarily have a causal relationship with the product. A serious AE is any AE that results in one of the following outcomes: death; life-threatening; requires in-patient hospitalization; results in a persistent or significant disability/incapacity; congenital anomaly/birth defect; other important medical event. The TEAEs are AEs that occur after the first dose of study treatment administration.
Time Frame: TEAEs were collected from the study drug administration (Day 1) up to end of the study, approximately 48 weeks.
Population: The Safety set included all subjects who received at least 1 dose of study treatment (EYP-1901 or sham).
Measure: Count of Participants; unit: Participants
Groups:
- Sham Injection - Study Eye; Sham Injection - Non-ocular: Subjects received a single dose of sham IVT injection on Day 1.
- Sham Injection - Non-study Eye; EYP-1901 2060 mcg - Non-study Eye; EYP-1901 3090 mcg - Non-study Eye: No study treatment administered in non-study eye.
- EYP-1901 2060 mcg - Study Eye; EYP-1901 2060 mcg - Non-ocular: Subjects received a single dose of EYP-1901 2060 mcg IVT injection on Day 1.
- EYP-1901 3090 mcg - Study Eye; EYP-1901 3090 mcg - Non-ocular: Subjects received a single dose of EYP-1901 3090 mcg IVT injection on Day 1.
Arm/Group | Sham Injection - Study Eye | Sham Injection - Non-study Eye | Sham Injection - Non-ocular | EYP-1901 2060 mcg - Study Eye | EYP-1901 2060 mcg - Non-study Eye | EYP-1901 2060 mcg - Non-ocular | EYP-1901 3090 mcg - Study Eye | EYP-1901 3090 mcg - Non-study Eye | EYP-1901 3090 mcg - Non-ocular
Number analyzed (Participants) | 26 | 26 | 26 | 26 | 26 | 26 | 25 | 25 | 25
Participants
  Any TEAE | 7 | 9 | 15 | 7 | 8 | 16 | 11 | 7 | 12
  Any Serious TEAE | 1 | 1 | 2 | 1 | 1 | 7 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: TEAEs were collected from the study drug administration (Day 1) up to end of the study, approximately 48 weeks.
Description: The Safety set included all subjects who received at least 1 dose of study treatment (EYP-1901 or sham).
Arm/Group | Sham Injection - Study Eye | Sham Injection - Non-study Eye | Sham Injection - Non-ocular | EYP-1901 2060 mcg - Study Eye | EYP-1901 2060 mcg - Non-study Eye | EYP-1901 2060 mcg - Non-ocular | EYP-1901 3090 mcg - Study Eye | EYP-1901 3090 mcg - Non-study Eye | EYP-1901 3090 mcg - Non-ocular
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26 | 1/26 | 0/26 | 0/26 | 1/26 | 0/25 | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 1/26 | 1/26 | 2/26 | 1/26 | 1/26 | 7/26 | 0/25 | 0/25 | 1/25
Other Adverse Events (participants affected / at risk) | 7/26 | 5/26 | 9/26 | 8/26 | 8/26 | 14/26 | 8/25 | 5/25 | 7/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham Injection - Study Eye (N=26) | Sham Injection - Non-study Eye (N=26) | Sham Injection - Non-ocular (N=26) | EYP-1901 2060 mcg - Study Eye (N=26) | EYP-1901 2060 mcg - Non-study Eye (N=26) | EYP-1901 2060 mcg - Non-ocular (N=26) | EYP-1901 3090 mcg - Study Eye (N=25) | EYP-1901 3090 mcg - Non-study Eye (N=25) | EYP-1901 3090 mcg - Non-ocular (N=25)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Diabetic retinopathy (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Macular oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endophthalmitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intraocular pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatic carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham Injection - Study Eye (N=26) | Sham Injection - Non-study Eye (N=26) | Sham Injection - Non-ocular (N=26) | EYP-1901 2060 mcg - Study Eye (N=26) | EYP-1901 2060 mcg - Non-study Eye (N=26) | EYP-1901 2060 mcg - Non-ocular (N=26) | EYP-1901 3090 mcg - Study Eye (N=25) | EYP-1901 3090 mcg - Non-study Eye (N=25) | EYP-1901 3090 mcg - Non-ocular (N=25)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic retinal oedema (Eye disorders) | 4 (4) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Diabetic retinopathy (Eye disorders) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Macular oedema (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Visual acuity reduced (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Glucose urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 2 (2)
Glycosylated haemoglobin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-03-31): https://cdn.clinicaltrials.gov/large-docs/09/NCT05383209/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-12): https://cdn.clinicaltrials.gov/large-docs/09/NCT05383209/SAP_001.pdf